CLINICAL TRIAL: NCT01283282
Title: Phase 4 Study of Clopidogrel in Patients With Stable Coronary Artery Disease to Determine Effects on Vascular Function, Biomarkers and Endothelial Progrenitor Cells
Brief Title: Investigation of the Athero-Protective Effects of Clopidogrel
Acronym: APECS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor of Medicine, Emory University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB00005145; APECS (Other: Other)
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Results first posted 2015-05-01 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clopidogrel/Placebo (Active Comparator): Subjects were randomized to clopidogrel 75 mg daily for 6 weeks. Then immediately transitioned to a placebo daily for 6 weeks.
  Interventions: Drug: Clopidogrel; Drug: Placebo
- Placebo/Clopidogrel (Active Comparator): Subjects were randomized to a placebo daily for 6 weeks. Then immediately transitioned to clopidogrel 75 mg daily for 6 weeks.
  Interventions: Drug: Clopidogrel; Drug: Placebo

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 75 mg PO qday for 6 weeks
  Other Names: Plavix
Drug: Placebo — Placebo PO qday for 6 weeks

SUMMARY:
The investigators would like to investigate whether clopidogrel will help lower the level of harmful markers in patients with coronary artery disease, and at the same time will help increase the cells that are useful in repairing the damaged blood vessels. The investigators will give half of the patients clopidogrel and the other half a sugar pill, placebo, and check the levels of these markers and helpful cells in each group. At the same time the investigators will check how well these patient's blood vessels work using ultrasound imaging of the forearm to see how blood vessels relax and tonometry to see how stiff the patient's blood vessels are. After 6 weeks of drug therapy, the patients will switch to the other drug and these same tests will be performed after an additional 6 weeks of therapy. The drug taken by the patient will not be known to the patient or the researchers. The patients will continue on their prescribed medical therapy during the duration of the 12 week study.

DETAILED DESCRIPTION:
Blockages in the blood vessels of the heart are caused by atherosclerosis. Atherosclerosis is the main cause for chest pain and heart attacks. Gradual narrowing of the vessels of the heart caused by blockages causes chronic symptoms, such as chest pain. Those with these findings often have a cardiac catheterization to detect these blockages. Additionally these patients may have an angioplasty or stent placed to help relieve these symptoms. With this angioplasty/stent procedure, patients are placed on the drug clopidogrel to help prevent clots from forming and narrowing of the blood vessels. Clopidogrel is a blood thinner that prevents clots from forming similar to an aspirin, but is more powerful and effective. Markers, or substances, have been identified that cause worsening of the blockages in the blood vessels of the heart. Many of these substances have been shown to decrease with the use of clopidogrel. This occurs separately from clopidogrel's ability to prevent clots. Endothelial progenitor cells, or EPCs, come mostly from the bone marrow and is helpful in repairing damage to the lining of the blood vessels of the heart. The EPCs help balance out the damage incurred in the blood vessels from those harmful markers. Several other drugs commonly used in heart disease have recently been shown to improve EPCs function. With this in mind, it is important to understand more of clopidogrel's function. A decrease in markers that cause worsening of the blockages, and an increase in the number of cells that will help repair damaged blood vessels of the heart is important in avoiding future chest pain and heart attacks. This may be how clopidogrel is currently protecting patients from developing new blockages. The investigators would like to investigate whether clopidogrel will help lower the level of harmful markers in patients with coronary artery disease, and at the same time will help increase the cells that are useful in repairing the damaged blood vessels. The investigators will give half of the patients clopidogrel and the other half a sugar pill, placebo, and check the levels of these markers and helpful cells in each group. At the same time the investigators will check how well these patient's blood vessels work using ultrasound imaging of the forearm to see how blood vessels relax and tonometry to see how stiff the patient's blood vessels are. After 6 weeks of drug therapy, the patients will switch to the other drug and these same tests will be performed after an additional 6 weeks of therapy. The drug taken by the patient will not be known to the patient or the researchers. The patients will continue on their prescribed medical therapy during the duration of the 12 week study.

ELIGIBILITY:
Inclusion Criteria:

* Male or females without child bearing potential aged 21-80 years
* Known coronary artery disease by angiogram or documented myocardial infarction.
* Able to provide written informed consent

Exclusion Criteria:

* Treated with clopidogrel or ticlodipine in the previous 3 months
* Age < 21 or >80 years
* Premenopausal females with potential for pregnancy
* Allergy to clopidogrel or aspirin
* Initiation or change in dose of any concomitant medical therapy within 2 months before the study
* Uncontrolled hypertension with BP>180 mmHg systolic and >120 mmHg diastolic
* Treated with coumadin therapy
* Intolerance or allergy to statins
* Acute infection in previous 4 weeks
* History of substance abuse
* Uninterpretable PAT test
* Current neoplasm
* Chronic renal failure [creatinine > 2.5 mg/dL] or liver failure (Liver enzymes >2X normal)
* Acute coronary syndrome, heart failure, CVA, coronary intervention within 3 months
* Known aortic stenosis, hypertrophic cardiomyopathy, symptomatic heart failure.
* Inability to give informed consent
* Inability to return to Emory for follow-up

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arshed A Quyyumi, MD, Principal Investigator — Emory University; Ziyad Ghazzal, MD, Principal Investigator — American University of Beirut, Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Ramadan R, Dhawan SS, Syed H, Pohlel FK, Binongo JN, Ghazzal ZB, Quyyumi AA. Effects of clopidogrel therapy on oxidative stress, inflammation, vascular function, and progenitor cells in stable coronary artery disease. J Cardiovasc Pharmacol. 2014 Apr;63(4):369-74. doi: 10.1097/FJC.0000000000000057. PMID 24336012

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from clinic sites at Emory University Hospital, Crawford Long Hospital, Grady Memorial Hospital and VA Medical Center between January 2008 through December 2008.
Groups:
- Placebo First/Then Clopidogrel: The subjects received placebo PO qd for the first 6 weeks then were switched to clopidogrel 75 mg PO qd therapy for an additional 6 weeks without any wash out period in between.
- Clopidogrel First/Then Placebo: The subjects received clopidogrel 75 mg PO qd for the first 6 weeks then were switched to placebo PO qd therapy for an additional 6 weeks without any wash out period in between.
Period: First Intervention (6 Weeks)
Arm/Group | Placebo First/Then Clopidogrel | Clopidogrel First/Then Placebo
Started | 25 | 23
Completed | 22 | 19
Not Completed | 3 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 1 | 0
Period: Second Intervention (6 Weeks)
Arm/Group | Placebo First/Then Clopidogrel | Clopidogrel First/Then Placebo
Started | 22 | 19
Completed | 22 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 41 subjects completed the entire study.
Groups:
- All Subjects: The subjects received clopidogrel 75 mg or placebo PO qd for the first 6 weeks then were switched to receive either placebo or clopidogrel 75 mg PO qd therapy for an additional 6 weeks without any wash out period in between.
Arm/Group | All Subjects
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Flow-mediated Dilation (FMD)
Description: Flow-mediated dilation (FMD) collected by an ultrasound and is measured by the percent change in diameter of the brachial artery from baseline to 12 weeks.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Error); unit: percent change in diameter
Groups:
- Clopridogrel: The subjects received clopidogrel 75 mg PO qd for the first 6 weeks or received clopidogrel 75 mg PO qd for the last 6 weeks.
- Placebo: The subjects received placebo PO qd for the first 6 weeks or the subjects received placebo PO qd for the last 6 weeks.
Arm/Group | Clopridogrel | Placebo
Number analyzed (Participants) | 41 | 41
percent change in diameter | 4.89 (0.59) | 4.81 (0.59)

2. Primary Outcome: Nitroglycerin-mediated Vasodilation
Description: Nitroglycerin (NTG)-mediated vasodilation was measured after 0.4 mg of NTG was administered sublingually. Brachial artery images were obtained via ultrasound after three minutes of NTG administration. Measurements from the twelve frames will be averaged to calculate the percent change in diameter of the brachial artery from baseline to 12 weeks.
Time Frame: Baseline, Week 12
Measure: Mean (Standard Error); unit: percent change in diameter
Arm/Group | Clopridogrel | Placebo
Number analyzed (Participants) | 41 | 41
percent change in diameter | 19.31 (1.49) | 17.10 (1.51)

3. Primary Outcome: Endothelial Progenitor Cells (EPCs)
Description: The circulating progenitor-enriched population of cells was measured by the expression of surface antigens using direct flow cytometry for CD34+, CD34+/CD133+, CD34+/ VEGF2R+ and CD34+/CD133+/VEGF2R+
Time Frame: Week 12
Measure: Mean (Standard Error); unit: cells/µL
Groups:
- Clopidogrel: The subjects received clopidogrel 75 mg PO qd for the first 6 weeks or received clopidogrel 75 mg PO qd for the last 6 weeks.
Arm/Group | Clopidogrel | Placebo
Number analyzed (Participants) | 41 | 41
cells/µL
  CD34+ | 1.46 (0.16) | 1.54 (0.21)
  CD34+/133+ | 0.68 (0.07) | 0.75 (0.16)
  CD34+/VEGF2R+ | 0.08 (0.03) | 0.09 (0.02)
  CD34+/CD133+/VEGF2R+ | 0.03 (0.009) | 0.03 (0.008)

4. Secondary Outcome: Pulse Wave Velocity (PWV)
Description: PWV was measured between the carotid and femoral arteries using the SphygmoCor device. Pressure waveforms at the carotid and femoral arteries were acquired using EKG gating. Velocity (distance per time in seconds) was calculated using the foot-to-foot method and the distance between the sites was measured manually.
Time Frame: Week 12
Measure: Mean (Standard Error); unit: m/s
Arm/Group | Clopridogrel | Placebo
Number analyzed (Participants) | 41 | 41
m/s | 8.77 (0.45) | 9.044 (0.45)

5. Secondary Outcome: Oxidative Stress Markers
Description: Oxidative stress was measured by using liquid chromatography to collect plasma cystine, cysteine, gluthione, and oxidized glutathione levels.
Time Frame: Week 12
Measure: Mean (Standard Error); unit: µM
Arm/Group | Clopridogrel | Placebo
Number analyzed (Participants) | 41 | 41
µM
  Cystine | 105.25 (7.36) | 102.39 (7.29)
  Cysteine | 13.71 (0.90) | 14.75 (0.89)
  Glutathione | 1.52 (0.17) | 1.71 (0.17)
  Oxidized glutathione | 0.08 (0.06) | 0.19 (0.06)

6. Secondary Outcome: Inflammatory Marker High-sensitivity C-reactive Protein (hsCRP)
Description: High-sensitivity C-reactive protein (hsCRP) was measured. The hsCRP levels were measured by Dade Behring nephelometry.
Time Frame: Week 12
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Clopridogrel | Placebo
Number analyzed (Participants) | 41 | 41
mg/L | 5.98 (1.95) | 4.31 (1.95)

7. Secondary Outcome: Inflammatory Marker CD40 Ligand
Description: CD40 ligand levels were measured. The level of CD40 ligand were measured using the Flurokine MultiAnalyte profiling (MAP) Human Base Kit B.
Time Frame: Week 12
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Clopridogrel | Placebo
Number analyzed (Participants) | 41 | 41
pg/mL | 1202.21 (318.35) | 2169.32 (318.35)

ADVERSE EVENTS:
Groups:
- Clopidogrel; Placebo: The subjects received clopidogrel 75 mg or placebo PO qd for the first 6 weeks then were switched to receive either placebo or clopidogrel 75 mg PO qd therapy for an additional 6 weeks without any wash out period in between.
Arm/Group | Clopidogrel | Placebo
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48

LIMITATIONS AND CAVEATS:
Limited sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes